CLINICAL TRIAL: NCT02657486
Title: Pilot Study of BGJ398 in Non-Muscle-Invasive Urothelial Carcinoma of the Bladder
Brief Title: BGJ398 in Non-Muscle-Invasive Urothelial Carcinoma of the Bladder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-090
Record Dates: First submitted 2016-01-13; First posted 2016-01-15 (Estimated); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Bladder Cancer; Non-Muscle-Invasive Urothelial Carcinoma
Keywords: BGJ398; 15-090
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — infigratinib

ARMS (1):
- BGJ398 (Experimental): BGJ398 will be administered at a dose of 125 mg orally once daily on a three weeks on, one week off schedule.
  Interventions: Drug: BGJ398

INTERVENTIONS:
Drug: BGJ398

SUMMARY:
The purpose of this study is to study the activity and effects of BGJ398 on bladder cancer tumors that are confined to the lining of the bladder.

ELIGIBILITY:
Inclusion Criteria:

* Recurrent high-risk non-muscle-invasive bladder cancer after prior intravesical BCG therapy meeting all of the following criteria:
* Histologically documented diagnosis of urothelial carcinoma confirmed by the Department of Pathology at MSKCC.
* Documentation of activating FGFR3 mutation or gene fusion on an assay performed in a CLIA-certified laboratory.
* History of high-grade, non-muscle-invasive bladder cancer (NMIBC).
* Clinical evidence of high-grade, stage pTa NMIBC.
* Prior intravesical therapy with at least one induction course of BCG
* Multiple papillary lesions with at least one amenable to marker tumor study (≤1 cm, non-invasive; or could be partially resected to leave a non-invasive lesion ≤1 cm) OR solitary papillary lesion amenable to marker tumor study (≤1 cm, non-invasive)
* Patient must be willing to consent to MSKCC protocol 12-245 ("Tumor Genomic Profiling in Patients Evaluated for Targeted Cancer Therapy"
* Age 18 years or older.
* Patient must be willing and able to comply with scheduled visits, treatment plan, and laboratory tests.
* Patient must be able to swallow and retain oral medication.
* Karnofsky performance status of ≥80.
* Recovery from adverse events of previous systemic anti-cancer therapies to baseline or grade 1, except for:

  * Alopecia
  * Stable neuropathy of ≤ grade 2 due to prior cancer therapy
* Women of childbearing potential, defined as all women physiologically capable of becoming pregnant, must agree to use highly effective methods of contraception during dosing and for 3 months following the discontinuation of study treatment.

Highly effective contraception methods include:

* Total abstinence (when this is in line with the preferred and usual lifestyle of the subject). Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.
* Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy) or tubal ligation at least six weeks before study treatment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow-up hormone level assessment.
* Male sterilization (at least 6 months prior to screening). For female subjects the vasectomized male partner should be the sole partner.
* Combination of any two of the following (a+b, a+c, or b+c):

  1. Use of oral, injected or implanted hormonal methods of contraception or other forms of hormonal contraception that have comparable efficacy (failure rate <1%); for example, hormone vaginal ring or transdermal hormone contraception.
  2. Placement of an intrauterine device (IUD) or intrauterine system (IUS)
  3. Barrier methods of contraception: Condom or Occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/vaginal suppository.

Oral contraceptives (OC), injected or implanted hormonal methods are not allowed as the sole method of contraception because BGJ398 has not been characterized with respect to the potential to interfere with PK and/or the effectiveness of OCs.

* If a woman is of non-childbearing potential, she must either:

  * Be post-menopausal as defined by 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms), OR
  * Have had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least six weeks ago. In the case of oophorectomy alone, the reproductive status of the woman must be confirmed by follow-up hormone level assessment.
* Sexually active males must use a condom during intercourse while taking drug and for three months after the last dose of the study drug. They should not father a child during this period. Men who have undergone vasectomy are also required to use a condom during intercourse to prevent delivery of the drug via seminal fluid.

Exclusion Criteria:

* Clinical suspicion of active CIS.
* Evidence of >1 area of CIS not associated with papillary tumor at this time.
* Evidence of >7 tumors present in the bladder.
* History or evidence of advanced urothelial carcinoma, including enlarged lymph nodes and/or distant metastases.
* Evidence of upper tract urothelial carcinoma.
* History of another primary malignancy within the last 3 years except:

  * Adequately treated in situ carcinoma of the cervix
  * Non-melanoma carcinoma of the skin
  * Any other curatively treated malignancy that has not been treated in the prior 3 months and is not expected to require treatment for recurrence during the course of the study.
* Patients who received prior treatment with a selective FGFR inhibitor.
* Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of oral BGJ398 (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, small bowel resection).
* History and/or current evidence of tissue calcification including, but not limited to, the soft tissue, kidneys, intestine, myocardium, and lung with the exception of calcified lymph nodes and asymptomatic vascular calcification.
* Current evidence of endocrine alterations of calcium/phosphate homeostasis, e.g., parathyroid disorders, history of parathyroidectomy, tumor lysis, tumoral calcinosis, etc.
* Use of medications that increase serum levels of phosphorus and/or calcium (e.g., calcium, phosphate, vitamin D, parathyroid hormone;) .
* Current evidence of corneal or retinal disorder/keratopathy including, but not limited to, bullous/band keratopathy, corneal abrasion, inflammation/ulceration, and/or keratoconjunctivitis, confirmed by ophthalmologic examination
* Treatment with any of the following anti-cancer therapies prior to the first dose of BGJ398 within the stated timeframes:

  * Cyclical chemotherapy (intravenous) within a period of time that is shorter than the cycle length used for that treatment (e.g., 6 weeks for nitrosourea, mitomycin-C).
  * Biological therapy (e.g., antibodies - including bevacizumab) within a period of time that is ≤ 5 half-lives or ≤ 4 weeks, whichever is shorter, prior to starting study drug.
  * Continuous or intermittent small molecule therapeutics within a period of time that is ≤ 5 half-lives or ≤ 4 weeks (whichever is shorter) prior to starting study drug.
  * Any other investigational agents within a period of time that is ≤ 5 half-lives or less than the cycle length used for that treatment or ≤ 4 weeks (whichever is shortest) prior to starting study drug.
  * Wide field radiotherapy (including therapeutic radioisotopes such as strontium 89) ≤ 4 weeks or limited field radiation for palliation ≤ 2 weeks prior to starting study drug.
* Patients who are currently receiving treatment with agents that are known strong inducers or inhibitors of CYP3A4
* Consumption of grapefruit, grapefruit juice, grapefruit hybrids, pomelos, pomegranates, star fruits, Seville oranges or related products within 7 days prior to first dose
* Use of herbal preparations/medications (including, but not limited to: St. John's wort, Kava, ephedra (ma huang), gingko bilboa, dehydroepiandrosterone (DHEA), yohimbe, saw palmetto, and ginseng within 7 days prior to first dose.
* Use of medications that are known to prolong the QT interval and/or are associated with a risk of Torsades de Pointes 7 days prior to first dose
* Use of amiodarone within 90 days prior to first dose
* Current use of therapeutic doses of warfarin sodium or any other coumadin-derivative anticoagulants. Heparin and/or low molecular weight heparins are allowed.
* Insufficient bone marrow function as evidenced by:

  * ANC <1,000/mm3 [1.0 x 10^9/L]
  * Platelets < 75,000/mm3 [75 x 10^9/L]
  * Hemoglobin < 10.0 g/dL
* Insufficient hepatic and renal function as evidenced by:

  * Total bilirubin > 1.5x ULN
  * AST/SGOT and ALT/SGPT > 2x ULN
  * Serum creatinine > 1.5x ULN
  * Calculated (using the CKD-EPI equation) or measured creatinine clearance < 75% LLN
* Calcium-phosphate homeostasis as evidenced by:

  * Inorganic Phosphorus outside of normal limits
  * Total serum calcium (can be corrected) outside of normal limits
* Clinically significant cardiac disease including any of the following:

  * Congestive heart failure requiring treatment (NYHA grade ≥ 2)
  * LVEF < 50 as determined by MUGA scan or ECHO
  * Uncontrolled hypertension (refer to WHO-ISH guidelines
  * History or presence of clinically significant ventricular arrhythmias, atrial fibrillation, resting bradycardia, or conduction abnormality
  * Unstable angina pectoris or acute myocardial infarction ≤ 3 months prior to starting study drug
  * QTcF > 480 msec (males and females)
  * History of congenital long QT syndrome
* Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the end of gestation, confirmed by a positive hCG laboratory test.
* Known positive serology for HIV, active Hepatitis B, and/or active Hepatitis C infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2016-01-06 (Actual); Primary Completion 2026-02-04 (Actual); Study Completion 2026-02-04 (Actual)

PRIMARY OUTCOMES:
tumor response | week 7
  with cystoscopy and cytology. A complete response will be defined as complete disappearance of the marker lesion at the week 7 evaluation, as determined by a negative cystoscopy and cytology.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Rosenberg, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/